CLINICAL TRIAL: NCT04636879
Title: Influence of Induced Expectations on the Autonomic Nervous System During a Dry Needling Intervention for Patients With Neck Pain. A Randomized Clinical Trial.
Brief Title: Dry Needling and Patients Treatment Expectations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, PhD. Daniel Pecos Martín, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI20/009
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain; Dry Needling; Motivation
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group 1. Positive expectation (Experimental): "Dry needling is a very effective tool used in the treatment of nonspecific neck pain, which we hope will reduce your neck pain."
  Interventions: Other: Positive expectation AND dry needling in the upper trapezius fibers, at the most painful point
- • Group 2. Neutral Expectation (Active Comparator): "Dry needling is an indicated tool used in the treatment of nonspecific neck pain, but its efficacy is unknown".
  Interventions: Other: Neutral expectation AND dry needling in the upper trapezius fibers, at the most painful point
- • Group 3. Negative Expectation (Active Comparator): "Dry needling is not a very effective treatment tool for nonspecific neck pain, so we expect your neck pain to increase a bit."
  Interventions: Other: Negative expectation AND dry needling in the upper trapezius fibers, at the most painful point

INTERVENTIONS:
Other: Positive expectation AND dry needling in the upper trapezius fibers, at the most painful point — The subjects will received the same treatment, using dry needling in the upper trapezius fibers, at the most painful point after receiving the corresponding message.
  Arms: • Group 1. Positive expectation
Other: Neutral expectation AND dry needling in the upper trapezius fibers, at the most painful point — The subjects will received the same treatment, using dry needling in the upper trapezius fibers, at the most painful point after receiving the corresponding
  Arms: • Group 2. Neutral Expectation
Other: Negative expectation AND dry needling in the upper trapezius fibers, at the most painful point — The subjects will received the same treatment, using dry needling in the upper trapezius fibers, at the most painful point after receiving the corresponding
  Arms: • Group 3. Negative Expectation

SUMMARY:
Objectives The aim of this study is to compare the effects of inducing positive expectations against negative or neutral induced expectations on the activation of the Autonomic Nervous System and the analgesic response, after a dry needling technique in upper trapezius fibers in patients with unspecific neck pain.

Summary Theoretical framework: Dry needling has proven its efficacy for the treatment of myofascial trigger points. Moreover, it has proven its effects over the Central Nervous System and the Autonomic Nervous System (ANS). Despite that previous studies have researched the role of patient's expectations and their relationship with the results of treatment, there is insufficient information concerning the effects of inducing expectations and the activation of the ANS during the application of widely used therapies, such as dry needling.

DETAILED DESCRIPTION:
The aim of this study will be to research the effects of induced expectations combined with a dry needling technique on the activation of the ANS and on the results of the treatment.

Hypothesis: The induction of a positive expectation shall cause a greater analgesic response associated with a response in the ANS compared to the induction of neutral or negative expectations.

Methods: Patients with neck pain will participated in this randomized clinical trial, which will be randomly assigned into 3 groups in order to receive positive, neutral or negative expectations concerning the treatment, by means of an individual informative talk. All subjects will received treatment using dry needling in the upper trapezius fibers. The main variables measured will be the following: Analogic Visual Scale, Pressure Pain Threshold using a mechanical Force Gage (before and after) and the activation of the ANS measuring the skin conductance, skin temperature, heart rate and breathing rate (monitored for 5 minutes before the intervention, during and 20 minutes afterwards).

ELIGIBILITY:
Inclusion Criteria:

* Neck pain.
* Hiperalgesic point in Upper trapezius muscle.

Exclusion Criteria:

* Pain Irradiation toward upper limb
* Psychological disorders
* Whiplash.
* Neuropathic symptoms
* Cervical and / or Shoulder Spine Surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Skin conductance (µS). | Change from baseline at twenty minutes
  It is the measure of the variations in the electrical resistance of the skin, caused by the excitation of the sweat glands, controlled by the Sympathetic Nervous System (SNS)

SECONDARY OUTCOMES:
Heart rate variability | Change from baseline at twenty minutes
  This variable is defined as the variation of the heartbeat in a previously defined period in an analysis of consecutive circadian periods. It measures the time in milliseconds between the R waves of two consecutive beats (known as the RR interval) and is widely used in the field of Cardiology for the stratification of patients after an acute myocardial infarction. It has also been shown to be a useful tool in detecting ANS activation.
Pain intensity | Change from baseline at twenty minutes
  It will be collected through the Visual Analogue Scale (VAS). It is a continuous scale, which consists of a 100 mm horizontal straight line, so that zero is equivalent to "total absence of pain" and 100 to "more bearable pain.
Pressure pain threshold | Change from baseline at twenty minutes.
  The pressure pain threshold is defined as the minimum amount of pressure necessary to cause pain. It has been measured through a Force Dial FDK using a mechanical Force Gage (Wagner Instruments).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Chair — Alcala University
Locations (1):
- Clinical University, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No